CLINICAL TRIAL: NCT06238167
Title: A Single Arm, Phase 2 Clinical Study Evaluating the Efficacy and Safety of Tislelizumab Plus Chemotherapy as Postoperative Adjuvant Therapy in Elderly Patients With Locally Advanced Gastric or Gastroesophageal Junction Adenocarcinoma
Brief Title: Tislelizumab Plus Chemotherapy as Postoperative Adjuvant Therapy in Elderly Patients With LA GC/GEJC
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: First Affiliated Hospital of Wenzhou Medical University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Bailu-D2-01
Record Dates: First submitted 2024-01-17; First posted 2024-02-02 (Actual); Last update posted 2024-02-02 (Actual); Status verified 2024-02

CONDITIONS: Gastric Cancer
Keywords: adjuvant therapy; elderly patients; tislelizumab; chemotherapy
MeSH Terms: conditions — Stomach Neoplasms | interventions — tislelizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Arm A (Experimental): Treatment arm(Tislelizumab+S-1/SOX)
  Enrolled patients will receive chemotherapy combined with tislelizumab postoperative adjuvant therapy. Chemotherapy regimens were determined by the investigator as S-1 therapy or low dose SOX therapy
  Interventions: Drug: Tislelizumab; Drug: S-1 therapy; Drug: low dose SOX therapy

INTERVENTIONS:
Drug: Tislelizumab — Tislelizumab, 200mg Q3W, max 16 cycles.
Drug: S-1 therapy — S1 d1-14 bid (< 1.25m^2 40mg, 1.25m^2-1.5m^2 50mg, ≥ 1.5m^2 60mg), followed by 7 days off (Q3W, max 16 cycles).
Drug: low dose SOX therapy — Oxaliplatin: 78mg/m^2, d1, S-1: 50mg d1-14 bid, followed by 7 days off (Q3W, max 8 cycles).

SUMMARY:
The purpose of study is to evaluate the efficacy and safety of postoperative adjuvant chemotherapy with tislelizumab in combination with tegafur-gimeracil-oteracil potassium (S-1 therapy) or tegafur-gimeracil-oteracil potassium + oxaliplatin (SOX therapy) in PD-L1 CPS positive, elderly (≥70years old), pStage III gastric cancer (including esophagogastric junction cancer) after D2 dissection.

DETAILED DESCRIPTION:
This is a prospective single-arm study to explore the safety and tolerability of chemotherapy combined with tislelizumab as postoperative adjuvant therapy in PD-L1 CPS positive, elderly, stage III gastric cancer/gastroesophageal junction adenocarcinoma.

Enrolled patients will receive chemotherapy combined with tislelizumab postoperative adjuvant therapy. Chemotherapy regimens were determined by the investigator as S-1 therapy or low dose SOX therapy:

S-1 therapy: S1 d1-14 bid (< 1.25m^ 40mg, 1.25m^2-1.5m2 50mg, ≥ 1.5m^2 60mg), followed by 7 days off (Q3W, max 16 cycles).

SOX treatment: oxaliplatin: 78mg/m2, d1, S-1: 50mg d1-14 bid, followed by 7 days off (Q3W, max 8 cycles).

Immunotherapy: Tislelizumab, 200mg Q3W, max 16 cycles.

The Primary endpoint is 1-year disease-free survival rate.

The secondary endpoints included:

1. 2-year disease-free survival rate, 3-year disease-free survival rate.
2. 2-year overall survival rate, 3-year overall survival rate.
3. Median disease-free survival
4. Median overall survival
5. Safety

ELIGIBILITY:
Inclusion Criteria:

* Patients with histologically confirmed adenocarcinoma of the stomach;
* Patients without a remnant cancer (R0) who have undergone gastrectomy within 6 weeks;
* According to the overall postoperative outcome, gastric cancer of stage III was determined according to the AJCC / UICC TNM Staging VII;
* Eastern Cooperative Oncology Group (ECOG) Performance Status (PS) score of 0 or 1;
* Patient with a confirmed pathological report related to the disease;
* No prior antitumor therapy (including immunotherapy, chemotherapy; radiotherapy), except for initial gastrectomy for primary lesions;
* PD-L1 CPS (22C3) score ≥1 ;
* Hematological examination: no obvious signs of hematological diseases: neutrophil count (ANC) ≥1.5×10^9/L, platelet count ≥100×10^9/L, hemoglobin ≥9 g/dL or ≥5.6 mmol/L, white blood cells ≥3.0×10^9/L, and no tendency to appear;Patients whose hematological indexes were at a critical value and could not meet the above criteria were determined by the researchers according to their physical conditions;
* Liver function test: alanine aminotransferase (ALT), aspartate aminotransferase (AST), alkaline phosphatase (ALP) ≤2.5×ULN, serum total bilirubin ≤1.5×ULN.For patients with Gilbert syndrome, serum total bilirubin < 3×ULN is required;
* Renal function test: serum creatinine (Cr) ≤1.5×ULN or creatinine clearance > 60ml/min (calculated according to Cockcroft-Gault).

Exclusion Criteria:

* Treatment with any other investigational drug or participation in another clinical trial with therapeutic intent within 28 days prior to enrollment;
* Postoperative complications that require clinical intervention and affect treatment, such as gastroparesis and dumping syndrome;
* Patients who are known to be allergic to or unable to tolerate the investigational drug;
* Uncontrolled serious medical conditions that the investigator believes will affect the subject's acceptance of the study protocol, such as co-existing serious medical conditions, including serious heart disease (such as New York Heart Association (NYHA) Class II or greater congestive heart failure), cerebrovascular disease, uncontrolled diabetes, uncontrolled hypertension, uncontrolled infections, etc.
* Known active HIV infection : untreated active HBV (defined as HBsAg positive with HBV-DNA copy number greater than the upper limit of normal in the laboratory of the study center) and HCV infection (HCV antibody positive with HCV-RNA level higher than the lower limit of detection);

Note: Hepatitis B subjects who meet the following criteria can also be enrolled:

1. HBV viral load <1000 copies /ml(20IU/ml) prior to initial dosing, subjects should receive anti-HBV therapy throughout study drug treatment to avoid viral reactivation;
2. For subjects with anti-HBC (+), HBsAg(-), anti-HBS (-) and HBV viral load (-), prophylactic anti-HBV therapy is not required, but close monitoring of viral reactivation is required;

   * Patients with malignant tumors other than gastric cancer (other than current gastric cancer) within the previous 5 years, patients will be eligible if all of the following criteria are met: treatment of malignant tumors for curative purposes, such as adequately treated cervical carcinoma in situ, non-melanoma skin cancer, localized prostate cancer after radical surgery (PSA≤10ng/ml);At the same time, according to the imaging follow-up results and any disease-specific tumor markers, no recurrence or metastasis was found.
   * ≥ Grade 2 (according to CTC AE v5.0) dysphagia, complete or incomplete gastrointestinal obstruction, active gastrointestinal bleeding, and perforation;
   * Patients who were judged by the investigator to be unsuitable for this study.

Min Age: 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2024-04-01 (Estimated); Primary Completion 2026-12-31 (Estimated); Study Completion 2028-12-31 (Estimated)

PRIMARY OUTCOMES:
1-year Disease-free survival rate | 1 year

SECONDARY OUTCOMES:
2-year Disease-free survival rate | 2 years
3-year Disease-free survival rate | 3 years
2-year overall survival rate | 2 years
3-year overall survival rate | 3 years
DFS | 3 years
OS | 3 years
Safety will be analyzed through the incidence of adverse events, serious adverse events | Up to 28 days from last dose

IPD SHARING:
Plan to Share IPD: No